CLINICAL TRIAL: NCT01886885
Title: The Efficacy of Mindfulness-Based Chronic Pain Management: A Pilot Study
Brief Title: Mindfulness Based Chronic Pain Management: A Pilot Study
Acronym: MBCPM
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: IRB_00061111
Record Dates: First submitted 2013-02-05; First posted 2013-06-26 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2013-06

CONDITIONS: Chronic Pain
Keywords: Mindfulness; Meditation; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MBCPM: There is just one group of participants of no more than 20 people.
  Interventions: Behavioral: Mindfulness Based Chronic Pain Management Intervention

INTERVENTIONS:
Behavioral: Mindfulness Based Chronic Pain Management Intervention — Mindfulness-Based Chronic Pain Management (MBCPM) is an intervention developed by Jackie Gardner-Nix, MD for individuals suffering from chronic pain. The focus of MBCPM is to teach clients skills that will facilitate the development of detached observation and reduce the experience of suffering through cognitive re-appraisal. The activities used within MBCPM include mindfulness meditation, gentle stretching/mindful movement, guided imagery, art techniques, psychoeducation, and discussion. There are daily homework assignments of just 5-30 minutes a day in MBCPM. Each class is two hours long with a break in the middle.

SUMMARY:
The primary objective for this pilot study is to determine if the Mindfulness-Based Chronic Pain Management (MBCPM) intervention would decrease pain and pain catastrophizing and increase pain acceptance in participants with chronic pain. The secondary objective is to explore if MBCPM will reduce depression and increase quality of life and mindfulness in the same group of participants. The additional aim of the pilot study is to evaluate the feasibility of conducting the MBCPM intervention in participants with chronic pain. We hypothesize that participants with chronic pain will show relatively good compliance with completing the MBCPM protocol and will show increased satisfaction associated with improvement in pain-related and other psychosocial indicators of functioning.

DETAILED DESCRIPTION:
The Institute of Medicine in their recent report Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research states that: "Common chronic pain conditions affect at least 116 million U.S. adults at a cost of $560-635 billion annually in direct medical treatment costs and lost productivity." (IOM, 2011, p. 1) Pain is defined as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage." (IASP, 2011). This widely accepted definition suggests that there are multiple components in the experience of pain, namely physiological and psychological. Pain has been reported as the most frequently reported symptom in primary care, while chronic pain is reported to affect 20-30% of the population in Western Countries. (Verhaak et al, 1998). Individuals with chronic pain often report co-morbid depression, anxiety, decreased quality of life, activity restriction, and inability to work or engage in productive activities. The most frequently used therapies are pharmacotherapy and surgical interventions, both of which have limitations in their effectiveness and tolerability.

A pressing need exists to develop alternative therapeutic modalities for caring for people with chronic pain. Mindfulness-based programs have emerged as effective interventions for different types of health conditions. Mindfulness is defined as "paying attention ina particular way, on purpose, in the present moment, and, non-judgmentally." (Kabat-Zinn, 1990) Research studies into mindfulness-based interventions have increased exponentially in the last three decades, based on the pioneering work of Jon Kabat-Zinn who developed Mindfulness-Based Stress Reduction (MBSR) in 1979. MBSR is a structured group based psycho-educational intervention that is conducted over a period of 8 weeks, with two hour classes occurring weekly. Each class teaches several mindfulness meditation practices such as sitting meditation, walking meditation, mindful yoga, and body scan. Participants are asked to complete homework assignments 6 out of 7 days following each session; these homework assignments provide opportunities to further engage in these practices so that they become more habitual. An all-day retreat occurs between weeks 6 and 7, providing further opportunities to engage in mindfulness practices.

Mindfulness-Based Chronic Pain Management (MBCPM) is an intervention developed by Jackie Gardner-Nix, MD, adapted from the standard MBSR curriculum for individuals suffering from chronic pain. The focus of this intervention is to teach clients skills that will facilitate the development of detached observation and reduce the experience of suffering through cognitive re-appraisal (Garder-Nix, 2008). The adaptations made in the MBCPM curriculum were based on the needs of individuals suffering from chronic pain; they include: increasing sessions to a 13 week long curriculum, replacing the mindful yoga with more gentle stretches, allowing participants to sit, stand, lie down, or move during sessions, and shortened mindfulness meditation practices. Additional therapeutic activities are also introduced throughout the program such as guided imagery and visualization, art techniques, and information about food and sleep. The length of homework assignments is also shortened from the original one hour length in MBSR to just 5-30 minutes a day in MBCPM, and there is no all-day Saturday retreat. These adaptations were made based on observations of difficulty that participants had with the original MBSR curriculum (Gardner-Nix, 2009b). Each class is two hours long with a break in the middle.

The current literature on chronic pain suggests that existing treatments have limited utility for chronic pain sufferers. "Currently available treatments have limited effectiveness for most people with severe chronic pain. For many such individuals, pain management on a daily basis takes place outside any health care setting." (IOM, 2011, p. 13) This statement from the Institute of Medicine report underscores the reasons why people turn to complementary and alternative medicine therapies - because they are not getting adequate relief from existing more conventional treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* English speaking
* Agree to participate
* Chronic pain for 3 months or more

Exclusion Criteria:

* Not speaking English
* Cognitive impairment
* Not able to commit to 13 week intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are 18 years of age and older, English speaking, in chronic pain for 3 months or more,and willing to participate in the 13 sessions.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The primary objective for this pilot study is to determine if the Mindfulness-Based Chronic Pain Management (MBCPM) intervention would decrease pain and pain catastrophizing and increase pain acceptance in participants with chronic pain. | 6 months
  The following assessments will be administered at the start of the intervention, at the end of the 13 week intervention, and at three month follow-up: Numerical Pain Rating Scale, Chronic Pain Acceptance Questionnaire, and the Pain Catastrophizing Scale

SECONDARY OUTCOMES:
The secondary objective is to explore if MBCPM will reduce depression and increase quality of life and mindfulness in the same group of participants. | 6 months
  The following assessments will be administered at the start of the intervention, at the end of the 13 week intervention, and at three month follow-up: Center for Epidemiologic Studies Depression Scale, the Five Factor Mindfulness Scale - Short Form, and the Quality of Life Scale.

OTHER OUTCOMES:
The additional aim of the pilot study is to evaluate the feasibility of conducting the MBCPM intervention in participants with chronic pain. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States